CLINICAL TRIAL: NCT01821651
Title: Use of Standardized Diagnostic Imaging Data (Computertomography, Angiography, Echocardiography) for Image Fusion in the Hybrid Operating Room
Brief Title: Use of Standardized Diagnostic Imaging Data for Image Fusion in the Hybrid Operating Room
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: HOR-1
Record Dates: First submitted 2012-12-10; First posted 2013-04-01 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Heart Valve Diseases
Keywords: TAVI; MitraClip; image modality; echocardiography; angiography
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HeartNavigator (Experimental): Group with HeartNavigator-Software
  Interventions: Device: HeartNavigator
- Control (Active Comparator): Control-group without HeartNavigator-Software
  Interventions: Other: Control-group HN
- EchoNav (Experimental): Group with EchoNav-Software
  Interventions: Device: EchoNav
- Conrol (Active Comparator): Control-group without EchoNav-Software
  Interventions: Other: Control-Group EN

INTERVENTIONS:
Device: HeartNavigator — Procedure with software
  Other Names: HeartNavigator, procedure with software
  Arms: HeartNavigator
Device: EchoNav — Procedure with software
  Other Names: EchoNav, procedure with software
  Arms: EchoNav
Other: Control-Group EN — Procedure without software
  Other Names: Compare to EchoNav-group
  Arms: Conrol
Other: Control-group HN — Procedure without software
  Other Names: Compare to HeartNavigator-group
  Arms: Control

SUMMARY:
Objectives:

Goal of the study is to investigate the potential benefit that transcatheter interventions such as Transcatheter Aortic Valve Implantation (TAVI), MitraClip, Left Atrial Appendage Closure and catheter Ablation can gain from multimodal image fusion techniques as they are available in the Hybrid suite.

Both the HeartNavigator and the EchoNav aim at decreasing the exposure to radiation and contrast agent, to shorten the operation time (efficacy), and to increase the quality of care (safety).

This pilot study aims at observing these aims on a small patient population and a control group.

Number of Subjects:

140 patients total in 6 groups:

* MitraClip, Left Atrial Appendage Closure or catheter Ablation with EchoNav (20, lead-in stage).
* MitraClip randomized with EchoNav (25), MitraClip randomized without EchoNav (25).
* TAVI with HeartNavigator lead in (10)
* TAVI randomized with HeartNavigator (30), TAVI randomized without HeartNavigator (30).

DETAILED DESCRIPTION:
Medical Device:

HeartNavigator: System for preoperative image-based assessment of aortic root geometry, planning of transcatheter aortic valve implantation, and intraoperative C-Arm control.

EchoNav: System for intraoperative registration of 3D Echo images with X-ray fluoroscopy images.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients over 18 years of age.
* Ability and willingness to give informed consent.
* Indication for TAVI, MitraClip, catheter ablation or percutaneous closure of the left atrial appendage procedure performed in the hybrid OR suite.
* Recent good quality CTA (TAVI patients only, no CTA needed for EchoNav).

Exclusion criteria:

* Contraindications on ethical grounds,
* Women who are pregnant or breast feeding,
* Emergency cases,
* Contraindication or known hypersensitivity to contrast media which is unresponsive to pretreatment with steroids and antihistamines,
* Known renal insufficiency (GFR < 50 ml/min) and patient is not on chronic hemodialysis (TAVI patients only, no contrast agent is necessary during MitraClip and transseptal puncture),
* Contraindications for transesophageal Echo (EchoNav patients only, TAVI is possible without TEE and TEE is not needed for the HeartNavigator),
* Known or suspected drug or alcohol abuse,
* Enrollment into a clinical trial within last 4 weeks if overlapping enrolment is not explicitly approved by ethics committee for the two trials,
* Patient is unable or unwilling to cooperate with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Radiation Dose (mSv) administered to each patient | Day of intervention (day 1)
  At the end of the procedure the recorded radiation-dose is assessed.

SECONDARY OUTCOMES:
Duration of the intervention (minutes) | Day of intervention (day 1)
  At the end of the procedure the skin-to-skin-time is assessed.
Contrast agent dose (ml) | Day of intervention (day 1)
  At the end of the procedure the recorded contrast agent dose is assessed.
Increased quality of care (EchoNav group) | Discharge: 1 to 5 days after intervention
  Usually 1 to 5 days after intervention
Degree of Mitral Regurgitation (EchoNav group) | Discharge: 1 to 5 days after intervention
  Usually 1 to 5 days after intervention
Postinterventional transvalvular gradient | Up to 7 days after intervention
  Catheter-based direct measurement

CONTACTS AND LOCATIONS:
Overall Officials: Volkmar Falk, Prof MD, Principal Investigator — University Hospital Zurich, Division of Cardiovascular Surgery
Locations (1):
- University Hospital Zurich, Division of Cardiovascular Surgery, Zurich, Canton of Zurich, Switzerland